CLINICAL TRIAL: NCT02519985
Title: Repeatability and Reproducibility of Corneal and Anterior Segment Measurements by ArcScan Insight 100 Very High-frequency Digital Ultrasound
Brief Title: Repeatability and Reproducibility of the ArcScan Insight 100 VHF Digital Ultrasound
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices currently awaiting software updates
Sponsor: London Vision Clinic (Other)
Collaborators: Arcscan, Inc. (Industry)
Responsible Party: Principal Investigator, Dan Reinstein, Medical Director, London Vision Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LoVC-005
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Corneal Thickness Measurement; Epithelial Thickness Measurement; Anterior Eye Segment Measurements
Keywords: VHF digital ultrasound; Corneal thickness; Epithelial thickness; Angle diameter; Sulcus diameter; Anterior chamber depth; Repeatability; Reproducibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Repeatability and Reproducibility of ArcScan Insight 100 (Experimental): For repeatability and reproducibility in normal eyes (n=20):
  Firstly, 5 consecutive repeated ArcScan Insight 100 scans of the cornea and anterior segment will be performed by the first operator.
  After a break of about 30 minutes, 5 consecutive repeated ArcScan Insight 100 scans of the cornea and anterior segment will be performed by the second operator.
  For repeatability and reproducibility in eyes after laser refractive surgery (n=20):
  Firstly, 5 consecutive repeated ArcScan Insight 100 scans of the cornea will be performed by the first operator.
  After a break of about 30 minutes, 5 consecutive repeated ArcScan Insight 100 scans of the cornea will be performed by the second operator.
  Interventions: Device: ArcScan Insight 100 very high-frequency digital ultrasound

INTERVENTIONS:
Device: ArcScan Insight 100 very high-frequency digital ultrasound — The ArcScan Insight 100 VHF digital ultrasound scanner that can measure individual layers within the cornea with very high precision, as well as being able to image the interior of the eye including the chamber between the iris and the cornea, the lens and other structures behind the iris.
  The ArcScan Insight 100 device is a digital ultrasound scanner, meaning that it uses ultrasound waves to measure parameters of the eye. The Insight examination involves the patient sitting in front of the ultrasound unit and looking through a disposable goggle-like eyepiece at a light source. Warm sterile balanced saline solution (like natural tears) are used to fill the space between the light source and the eye, to allow ultrasound transmission. There is no contact between the instrument and the eye other than being immersed in this water bath.
  Other Names: VHF digital ultrasound

SUMMARY:
The purpose of this study is to evaluate the repeatability and reproducibility of corneal (including corneal, epithelial, stromal, and LASIK flap thickness) and anterior segment measurements using the ArcScan Insight 100 very high-frequency digital ultrasound arc-scanner.

DETAILED DESCRIPTION:
Very high-frequency (VHF) digital ultrasound was first used in 1993 to obtain images of the cornea (the window at the front of the eye) and anterior segment (the space behind the cornea including the iris and the lens). A commercially available instrument, called the Artemis 2, has been used in routine clinical practice since 2001. The Artemis 2 was CE approved as well as having FDA approval (the US equivalent of the CE mark).

The ArcScan Insight 100 VHF digital ultrasound scanner is a new instrument so does not yet have a CE mark. However, the ArcScan Insight 100 is an upgraded version of the Artemis 2, so any differences are improvements to components, but the measurement method remains essentially the same.

The aim of the study is to establish the repeatability (i.e. the variability in measurements taken by a single examiner during a single visit) and reproducibility (i.e. the variability in measurements taken in the same conditions between two examiners) of the ArcScan Insight 100 device for measuring corneal and anterior segment parameters.

ELIGIBILITY:
INCLUSION CRITERIA Only patients who are medically suitable for corneal refractive surgery can be included in the study.

As general inclusion criteria the following aspects are defined:

* Subjects should be 21 years of age or older.
* Contact lens wearers must stop wearing their contact lenses at least four weeks per decade of wear before baseline measurements in case of hard contact lenses and one week before baseline measurements in case of soft contact lenses.
* Patient will be able to understand the patient information and willing to sign an informed consent.

For the repeatability and reproducibility phase using normal eyes of the study:

* Eyes with no ocular pathology
* Eyes with no previous ocular or corneal surgery

For the repeatability and reproducibility phase using post-LASIK eyes of the study:

• Eyes between 3 and 9 months after LASIK or SMILE

For the comparison of ArcScan Insight 100 VHF digital ultrasound with RTVue OCT

• Either eyes before or after corneal refractive surgery

EXCLUSION CRITERIA

* Previous ocular or corneal surgery (for normal eyes)
* Patient not being able to tolerate local or topical anesthesia
* Patient has active conjunctivitis or any active ocular infection or inflammation
* Patient has a corneal ulcer
* Patient has an open wound on the corneal epithelium
* Patient has compromised epithelium (e.g. ≥Grade 3 superficial punctate keratitis)
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Repeatability of ArcScan Insight 100 corneal scans in normal eyes (standard deviation) | 1 day
  The standard deviation of 5 repeated measurements for corneal thickness, epithelial thickness, and stromal thickness in normal eyes with no previous corneal surgery

SECONDARY OUTCOMES:
Reproducibility of ArcScan Insight 100 corneal scans in normal eyes (between-operator standard deviation) | 1 day
  The between-operator standard deviation of 5 repeated measurements for each operator for corneal thickness, epithelial thickness, and stromal thickness in normal eyes with no previous corneal surgery
Repeatability of ArcScan Insight 100 anterior segment scans in normal eyes (standard deviation) | 1 day
  The standard deviation of 5 repeated measurements for anterior segment dimensions: angle diameter, sulcus diameter, anterior chamber depth, and lens rise from the zonular plane in normal eyes with no previous corneal surgery
Reproducibility of ArcScan Insight 100 anterior segment scans in normal eyes (between-operator standard deviation) | 1 day
  The between-operator standard deviation of 5 repeated measurements for each operator for anterior segment dimensions: angle diameter, sulcus diameter, anterior chamber depth, and lens rise from the zonular plane in normal eyes with no previous corneal surgery
Repeatability of ArcScan Insight 100 corneal scans in eyes after corneal laser refractive surgery (standard deviation) | 1 day
  The standard deviation of 5 repeated measurements for corneal thickness, epithelial thickness, stromal thickness, flap thickness, and residual stromal thickness in eyes after corneal laser refractive surgery
Reproducibility of ArcScan Insight 100 corneal scans in eyes after corneal laser refractive surgery (between-operator standard deviation) | 1 day
  The between-operator standard deviation of 5 repeated measurements for each operator for corneal thickness, epithelial thickness, stromal thickness, flap thickness, and residual stromal thickness in eyes after corneal laser refractive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dan Z Reinstein, MD MA, Principal Investigator — London Vision Clinic
Locations (1):
- London Vision Clinic, London, United Kingdom

REFERENCES:
- [Background] Reinstein DZ, Silverman RH, Raevsky T, Simoni GJ, Lloyd HO, Najafi DJ, Rondeau MJ, Coleman DJ. Arc-scanning very high-frequency digital ultrasound for 3D pachymetric mapping of the corneal epithelium and stroma in laser in situ keratomileusis. J Refract Surg. 2000 Jul-Aug;16(4):414-30. doi: 10.3928/1081-597X-20000701-04. PMID 10939721
- [Background] Paul T, Lim M, Starr CE, Lloyd HO, Coleman DJ, Silverman RH. Central corneal thickness measured by the Orbscan II system, contact ultrasound pachymetry, and the Artemis 2 system. J Cataract Refract Surg. 2008 Nov;34(11):1906-12. doi: 10.1016/j.jcrs.2008.07.013. PMID 19006737
- [Background] Ursea R, Feng M, Urs R, RoyChoudhury A, Silverman RH. Comparison of artemis 2 ultrasound and Visante optical coherence tomography corneal thickness profiles. J Refract Surg. 2013 Jan;29(1):36-41. doi: 10.3928/1081597X-20121126-01. Epub 2012 Nov 30. PMID 23205905
- [Background] Ogbuehi KC, Osuagwu UL. Repeatability and interobserver reproducibility of Artemis-2 high-frequency ultrasound in determination of human corneal thickness. Clin Ophthalmol. 2012;6:761-9. doi: 10.2147/OPTH.S31690. Epub 2012 May 21. PMID 22693418
- [Background] Pinero DP, Plaza AB, Alio JL. Anterior segment biometry with 2 imaging technologies: very-high-frequency ultrasound scanning versus optical coherence tomography. J Cataract Refract Surg. 2008 Jan;34(1):95-102. doi: 10.1016/j.jcrs.2007.08.033. PMID 18165088